CLINICAL TRIAL: NCT00061009
Title: Relationship of Autonomic Function to Hypnotic Susceptibility
Brief Title: Hypnosis in Autonomic Function
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030199; 03-N-0199
Record Dates: First submitted 2003-05-19; First posted 2003-05-20 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2006-01

CONDITIONS: Vasovagal Syncope; Postural Tachycardia Syndrome; Hypnosis
Keywords: Chronic Orthostatic Intolerance; Dysautonomia; Postural Tachycardia Syndrome; Neurocardiogenic; Syncope; Neurocardiogenic Syncope; COI; POTS; Neurocardogenic Syncope; NCS; Healthy Volunteer; HV
MeSH Terms: conditions — Syncope, Vasovagal; Postural Orthostatic Tachycardia Syndrome; Autonomic Nervous System Diseases; Syncope

SUMMARY:
This study will investigate the relationship between susceptibility to hypnosis and regulation of the autonomic nervous system (nerves that control involuntary body functions, such as heart rate and sweating).

Hypnosis is a state of mind in which the individual is highly focused, relatively unaware of his or her surroundings, and possibly more able to accept and use therapeutic suggestions. People vary in their responsiveness, or susceptibility, while in hypnosis. People with certain conditions, such as chronic fatigue syndrome (CFS), chronic pain, posttraumatic stress disorder (PTSD), and generalized anxiety disorder (GAD) have altered hypnotic susceptibility. Patients with chronic orthostatic intolerance (COI) often have symptoms similar to those of individuals with CFS, chronic pain, PTSD, and GAD, and this study will examine how patients with COI respond to hypnosis as compared with healthy normal volunteers. COI is a group of disorders characterized by intolerance to prolonged standing. Among them are neurocardiogenic syncope (NCS), in which patients have recurrent episodes of sudden loss of consciousness, and postural tachycardia syndrome (POTS), in which patients have a sustained increase in heart rate after standing.

In addition to the comparison of COI and normal volunteer responses to hypnosis, the study will examine how hypnotic susceptibility is related to the ability to control autonomic functions such as blood pressure, heart rate, and sweating. The autonomic nervous system is activated when the body is stressed, not only from physical stimuli such as cold temperature, but also from mental stimuli, such as seeing a rattlesnake up close. Hypnosis may, therefore, be a useful tool to understand how the mind controls the autonomic nervous system.

Healthy normal volunteers and patients with NCS or POTS who are 18 years of age or older may be eligible for this two-part study. In part 1, participants complete a questionnaire and are then tested for hypnotic susceptibility. For this test, a professionally trained physician guides the subject through a procedure to achieve a hypnotic state. The subject is asked to perform several simple tasks and is then guided back to a normal state of being. In part 2, the subject undergoes hypnosis again, during which the physician offers various suggestions while monitoring activity of the subject's autonomic nervous system. The subject is connected to various sensors that continuously monitor blood pressure, heart rate, blood flow, sweat response, skin electrical conduction, and brain wave activity. An intravenous catheter is inserted into an arm vein to collect blood samples. At the end, the subject is guided back to a normal state of being.

The hypnosis session in part 1 is videotaped in order to: 1) permit review by a scientist who is unaware of the subject's condition and whose judgment will not, therefore, be biased; and 2) have a record of the experimental data. Only qualified investigators will view the videotape.

DETAILED DESCRIPTION:
This protocol describes a study to investigate the relationship between susceptibility to hypnosis and regulation of the autonomic nervous system. Several studies have demonstrated that individuals with particular conditions such as chronic fatigue syndrome (CFS), posttraumatic stress disorder (PTSD), chronic pain, and generalized anxiety disorder (GAD), have altered hypnotic susceptibility. Patients with chronic orthostatic intolerance (COI), a general category of autonomic dysfunction that includes neurocardiogenic syncope (NCS) and postural tachycardia syndrome (POTS), often present with symptoms that are similar to those seen in CFS, PTSD, chronic pain, or GAD. These observations led to the hypothesis tested in this protocol that patients with COI may also have altered hypnotic susceptibility. We also hypothesize that increased hypnotic susceptibility will correlate with increased ability to modulate autonomic function appropriately in response to suggestions during hypnosis.

The study population includes normal volunteers and patients with NCS or POTS. The design is blinded and correlative. Primary outcome measures are hypnotic susceptibility as measured by standardized scales; self-report inventory scores of psychobehavioral variables; physiologic parameters such as hemodynamics, sweating, skin electrical conductance, body temperature, respiratory rate, and bispectral analysis; and plasma catechol levels. The results of this study may lead to novel therapeutic strategies using hypnosis for COI.

ELIGIBILITY:
INCLUSION CRITERIA:

Subjects are patients with COI (POTS or NCS) identified in existing diagnostic protocols of the Clinical Neurocardiology Section (CNCS) and age- and gender-matched healthy volunteers. Patients with COI must be evaluated first through these diagnostic protocols prior to being offered enrollment in this protocol. Participation in this protocol is offered to subjects independently of gender, race, ethnicity, religion, or creed.

The studies in this protocol can be performed on an outpatient basis. Inpatients may also participate as long as participation does not interfere with the protocol(s) under which they have been admitted.

EXCLUSION CRITERIA:

Subjects are excluded based on: age less than 18 years, unwillingness to be hypnotized or videotaped; religious or other beliefs that would prevent engagement in hypnosis; psychosis or psychotic depression; non-fluency in spoken English; and inability to participate adequately in the tasks of the hypnotic susceptibility scale. In addition, patients are excluded if they are being treated with, and cannot discontinue, a drug likely to interfere with the scientific results. An example would be treatment with a beta-adrenoceptor blocker. Patients unable to discontinue nicotine or alcohol temporarily are excluded. Patients are not to discontinue any medications before the patient or the patient's doctor discusses this with the Principal Investigator, or the Research Nurse. If it is decided that discontinuing medications would be unsafe, then the patient is excluded from the study. Finally, subjects are excluded if there are technical limitations in placing an i.v. or monitoring devices.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 93
Dates: Start 2003-05; Study Completion 2006-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Goldstein DS, Robertson D, Esler M, Straus SE, Eisenhofer G. Dysautonomias: clinical disorders of the autonomic nervous system. Ann Intern Med. 2002 Nov 5;137(9):753-63. doi: 10.7326/0003-4819-137-9-200211050-00011. PMID 12416949
- [Background] Goldstein DS, Holmes C, Frank SM, Naqibuddin M, Dendi R, Snader S, Calkins H. Sympathoadrenal imbalance before neurocardiogenic syncope. Am J Cardiol. 2003 Jan 1;91(1):53-8. doi: 10.1016/s0002-9149(02)02997-1. PMID 12505571
- [Background] Accurso V, Winnicki M, Shamsuzzaman AS, Wenzel A, Johnson AK, Somers VK. Predisposition to vasovagal syncope in subjects with blood/injury phobia. Circulation. 2001 Aug 21;104(8):903-7. doi: 10.1161/hc3301.094910. PMID 11514377